CLINICAL TRIAL: NCT02513992
Title: Early Ictal SPECT With Intra-arterial Injection to Localize the Ictal Onset Zone in Refractory Focal Epilepsy.
Brief Title: Ictal SPECT With Intra-arterial Injection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no patient met inclusion criteria
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr W Van Paesschen, Prof. Dr., Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S58243
Record Dates: First submitted 2015-07-19; First posted 2015-08-03 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Epilepsy
Keywords: ictal SPECT
MeSH Terms: conditions — Epilepsy | interventions — technetium Tc 99m bicisate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intra-arterial injection of tracer (Experimental): The perfusion tracer 99m-Technetium Ethyl Cysteinate Dimer will be injected via an intra-arterial catheter by a pressure injector to obtain a subtracted ictal SPECT co-registered with MRI (SISCOM)
  Interventions: Procedure: intra-arterial injection of tracer; Drug: 99m-Technetium Ethyl Cysteinate Dimer; Device: intra-arterial catheter; Device: pressure injector

INTERVENTIONS:
Procedure: intra-arterial injection of tracer — intra-arterial ictal injection of perfusion tracer
Drug: 99m-Technetium Ethyl Cysteinate Dimer — administration of perfusion tracer 99m Tc-ECD during epileptic seizure
  Other Names: 99m Tc-ECD
Device: intra-arterial catheter — placement of intra-arterial catheter via femoral artery
Device: pressure injector — the injection of the perfusion tracer will be delivered with a pressure injector

SUMMARY:
Ictal SPECT with intravenous injection in a cubital vein of a perfusion tracer is an established technique to localize the ictal onset zone during presurgical evaluation of refractory focal epilepsy. When seizures last less than 10 seconds, localizing information is often not obtained. Since it takes around 30 seconds before the tracer reaches the brain after intravenous injection, ictal hyperperfusion most likely has already switched to postictal hypoperfusion. In this study, we plan to inject the perfusion tracer in the aorta proximal to the cerebral arteries, which will allow a true ictal injection in patients with seizures of short duration.

DETAILED DESCRIPTION:
In this study, the investigators will select one patient with refractory focal epilepsy with frequent seizures of short duration, which can not be localized with early ictal SPECT with intravenous injection in a cubital vein. An arterial catheter will be inserted. The right groin will be disinfected using an alcoholic disinfectant and locally anaesthetized. The artery in the groin, the femoral artery, will be punctured. A catheter is inserted in the artery and slided towards the heart. To determine the correct position of the catheter proximal to the cerebral arteries, a contrast agent will be injected, and at the same time radiographs will be taken. The catheter will be attached and taped in the groin. The patient will be monitored with video-EEG recording. During an epileptic seizure, the perfusion tracer 99m-Technetium Ethyl Cysteinate Dimer (99mTc- ECD) dissolved in 30 cc normal saline will be injected with a pressure injector over 2 seconds. After injection, the catheter will be removed and the ictal SPECT scan will be performed. Subtracted ictal SPECT images co-registered with MRI (SISCOM) will be obtained. The investigators plan to do this study in one patient in order to assess whether this procedure is logistically possible and to determine whether subtraction images of ictal SPECT with intra-arterial injection minus interictal SPECT with intravenous injection allows localization of the ictal onset zone.

ELIGIBILITY:
Inclusion Criteria:

* Refractory unifocal epilepsy
* Early ictal SPECT with intravenous injection did not localize the ictal onset zone
* Several seizure per day, or clusters of several seizures per day
* Seizures are of short duration (i.e. less than 10-15 seconds)
* Patient asks for epilepsy surgery

Exclusion Criteria:

* Renal failure
* Allergy to contrast agents
* Fever
* Anemia
* Usage of anticoagulants
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Correct localization of the ictal onset zone | 1 year after epilepsy surgery
  seizure free outcome will be assessed 1 year after epilepsy surgery and correlated with Subtracted ictal SPECT co-registered with MRI (SISCOM) results

CONTACTS AND LOCATIONS:
Overall Officials: Wim Van Paesschen, MD PhD, Principal Investigator — UZ Leuven/KU Leuven
Locations (1):
- University Hospitals Leuven, department of Neurology, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Van Paesschen W, Dupont P, Van Driel G, Van Billoen H, Maes A. SPECT perfusion changes during complex partial seizures in patients with hippocampal sclerosis. Brain. 2003 May;126(Pt 5):1103-11. doi: 10.1093/brain/awg108. PMID 12690050
- [Background] Van Paesschen W. Ictal SPECT. Epilepsia. 2004;45 Suppl 4:35-40. doi: 10.1111/j.0013-9580.2004.04008.x. PMID 15281956
- [Background] Van Paesschen W, Dupont P, Sunaert S, Goffin K, Van Laere K. The use of SPECT and PET in routine clinical practice in epilepsy. Curr Opin Neurol. 2007 Apr;20(2):194-202. doi: 10.1097/WCO.0b013e328042baf6. PMID 17351491
- [Background] Goffin K, Dedeurwaerdere S, Van Laere K, Van Paesschen W. Neuronuclear assessment of patients with epilepsy. Semin Nucl Med. 2008 Jul;38(4):227-39. doi: 10.1053/j.semnuclmed.2008.02.004. PMID 18514079
- [Background] Tousseyn S, Dupont P, Goffin K, Sunaert S, Van Paesschen W. Correspondence between large-scale ictal and interictal epileptic networks revealed by single photon emission computed tomography (SPECT) and electroencephalography (EEG)-functional magnetic resonance imaging (fMRI). Epilepsia. 2015 Mar;56(3):382-92. doi: 10.1111/epi.12910. Epub 2015 Jan 29. PMID 25631544
- [Background] Cleeren E, Casteels C, Goffin K, Janssen P, Van Paesschen W. Ictal perfusion changes associated with seizure progression in the amygdala kindling model in the rhesus monkey. Epilepsia. 2015 Sep;56(9):1366-75. doi: 10.1111/epi.13077. Epub 2015 Jul 15. PMID 26174547